CLINICAL TRIAL: NCT03142516
Title: A Phase II Trial to Evaluate the Efficacy and Safety of FOLFIRI + Panitumumab as First-line Treatment in Elderly Patients With RAS/BRAF Wild-type Unresectable Metastatic Colorectal Cancer and Good Performance Status
Brief Title: FOLFIRI + Panitumumab First-line Treatment in Elderly Patients With Unresectable Metastatic Colorectal Cancer, RAS/BRAF Wild-type and Good Performance Status
Acronym: OPALO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol Multidisciplinario del Cancer Digestivo (Other)
Collaborators: Amgen (Industry); Pivotal S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEMCAD-16-03; 2017-001639-38 (EudraCT Number)
Record Dates: First submitted 2017-05-02; First posted 2017-05-05 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Colorectal Neoplasms; Colorectal Carcinoma; Colorectal Cancer Metastatic; Neoplasm Metastasis
Keywords: Clinical Trial, Phase II; Elderly; Aged; Disease-Free Survival; Safety; Tolerability; Chemotherapy regimen; Monoclonal antibody; FOLFIRI; Panitumumab; RAS/BRAF Wild-type
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Panitumumab; Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FOLFIRI + panitumumab (Experimental): All patients will receive panitumumab plus FOLFIRI for disease control in 14-day cycles until disease progression, unacceptable toxicity, investigator's decision or patient withdrawal of consent, at the following doses:
  * Panitumumab: 6 mg/kg administered by intravenous (IV) infusion over 60 min on days 1 and 14 of every cycle just before administration of chemotherapy
  * FOLFIRI
  * Irinotecan: 150 mg/m2 as IV infusion over 90 min on day 1of first treatment cycle. If tolerance of this first dose is good, it will be scaled to a full dose of 180 mg/m2 starting from the second treatment cycle.
  * Folinic acid: (leucovorin) 200-400 mg/m2 IV over 2 hours on day 1
  * 5-FU: 400 mg/m2 bolus followed by 2400 mg/m2 IV continuous infusion over 46-48 hours on days 1 and 2
  Interventions: Drug: Panitumumab; Drug: Irinotecan; Drug: Folinic acid; Drug: 5-FU

INTERVENTIONS:
Drug: Panitumumab — Panitumumab 6 mg/kg will be administered by intravenous (IV) infusion over 60 min on days 1 and 14 of every cycle just before administration of chemotherapy
  Other Names: Vectibix
Drug: Irinotecan — Irinotecan 150 mg/m2 will be administered as IV infusion over 90 min on day 1of first treatment cycle. If tolerance of this first dose is good, it will be scaled to a full dose of 180 mg/m2 starting from the second treatment cycle
  Other Names: Any marketed
Drug: Folinic acid — Folinic acid 200-400 mg/m2 will be administered as IV infusion over 2 hours on day 1
  Other Names: Leucovorin; Any marketed
Drug: 5-FU — 5-FU will be administered IV 400 mg/m2 bolus followed by 2400 mg/m2 IV continuous infusion over 46-48 hours on days 1 and 2
  Other Names: 5-fluorouracil; Any marketed

SUMMARY:
To estimate progression-free survival at one year in elderly patients with RAS/BRAF wild-type unresectable mCRC and good performance status treated with FOLFIRI + panitumumab as first-line therapy.

The clinical hypothesis of this study is that the combination of panitumumab and FOLFIRI is a good treatment option in elderly patients with good performance status and RAS/BRAF wild-type unresectable mCRC. Another purpose of this clinical trial is to determine the RAS/BRAF mutation status in liquid biopsies at baseline and at the time of disease progression.

DETAILED DESCRIPTION:
Phase II, multicentre, single-arm trial. Elderly patients with good performance status and RAS/BRAF wild-type unresectable mCRC will be evaluated before being included in this trial. Eligible patients will receive panitumumab plus FOLFIRI for disease control until disease progression, unacceptable toxicity, investigator decision or the patient's withdrawal of consent.

Tumour response will be evaluated by investigators using RECIST criteria (Response Evaluation Criteria in Solid Tumours) version 1.1. Tumour response will be evaluated every 8 weeks until disease progression is documented. Disease response will be confirmed no less than 28 days after the criteria for response are first met. Radiographic progression of subjects with symptoms indicating disease progression will be evaluated at the time of symptom onset.

Following disease progression, information will be collected on the subsequent lines of treatment chosen by the investigator and survival at follow-up visits held every 12 weeks (± 4 weeks) until completion of the trial (approximately 24 months after inclusion of the last patient in the trial).

A blood sample will be taken at baseline and at the time of disease progression in order to determine the RAS/BRAF mutation status.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 70 years,
2. Able to understand, sign and date an informed consent form approved by the IEC,
3. Histologically confirmed colorectal carcinoma with metastatic disease,
4. RAS/BRAF wild-type status in solid biopsy confirmed prior to inclusion of the study,
5. No previous treatment for metastatic disease,
6. Patients starting therapy with FOLFIRI + panitumumab with a treatment aim other than achieving potential resectability of the disease,
7. Independence in activities of daily living (ADL) based on the Katz Index and in instrumental activities of daily living (IAL) based on the Lawton Index,
8. Having no or only one comorbidity according to the Charlson Comorbidity Index. The following ones are not considered comorbidities as long as it is provided they are adequately controlled with medication: gastroduodenal ulcer, diabetes without target organs' damage, chronic respiratory disease and connective tissue disease.
9. Presence of at least one unidimensional measurable lesion ≥ 10 mm according to RECIST criteria (version 1.1),
10. ECOG (Eastern Cooperative Oncology Group) performance status of 0-1,
11. Adequate bone marrow function: neutrophils ≥ 1.5 x 10^9/l; platelets ≥ 100 x 10^9/l; haemoglobin ≥ 9 g/dl,
12. Hepatic, renal and metabolic function as follows:

    1. Total bilirubin count ≤ 1.5 x ULN; ALT and AST < 5 x ULN;
    2. Renal function, calculated creatinine clearance or 24-hour creatinine clearance ≥ 50 ml/min;
    3. Magnesium > LLN

Exclusion Criteria:

1. Diagnosed or suspected central nervous system (CNS) metastasis,
2. Patients with initially resectable metastases at the time of diagnosis of metastatic disease.
3. History or presence of another malignancy, with the exception of curatively treated in situ carcinoma of the cervix or non-melanoma skin cancer or any curatively treated solid tumour, with no active disease or administration of treatment within 5 years prior to inclusion in the study,
4. Prior treatment with irinotecan,
5. Prior adjuvant chemotherapy for colorectal cancer terminated less than 6 months before metastatic disease was diagnosed,
6. Prior anti-epidermal growth factor receptor (EGFR) antibody therapy (eg, cetuximab), anti- vascular endothelial growth factor (VEGF) or treatment with small molecule EGFR inhibitors (eg, erlotinib),
7. Unresolved toxicities from prior systemic treatment that, in the investigator's opinion, make the patient unsuitable for inclusion,
8. Hormone therapy, immunotherapy with experimental or approved antibodies/proteins (e.g. bevacizumab) ≤ 30 days prior to inclusion,
9. Evidence of previous acute hypersensitivity reaction of any grade to any of the components of the treatment,
10. History of interstitial lung disease or pulmonary fibrosis or signs of interstitial lung disease or pulmonary fibrosis on baseline CT,
11. Presence of geriatric syndromes, defined as dementia, repeated falls, fecal incontinence or urinary incontinence,
12. Acute or subacute bowel obstruction and/or active bowel disease or another bowel disease causing chronic diarrhoea (defined as diarrhoea of grade ≥ 2 according to the NCI (National Cancer Institute) Common Terminology Criteria for Adverse Events (CTCAE version 4.03),
13. Significant cardiovascular disease, including unstable angina pectoris or myocardial infarction within 12 months prior to inclusion in the study,
14. History of Gilbert's syndrome or dihydropyrimidine dehydrogenase deficiency,
15. Positive test result for human immunodeficiency virus, hepatitis C virus, chronic active hepatitis B infection,
16. Treatment for systemic infection within 14 days prior to the start of the study treatment,
17. Clinically significant sensory peripheral neuropathy,
18. Any concurrent disease that may increase the risk associated with study participation or may interfere with the interpretation of study results,
19. Any investigational product within 30 days prior to inclusion,
20. Surgery (not including diagnostic biopsy or the placement of a central line) and/or radiotherapy within 28 days prior to inclusion in the study,
21. Males whose partner is of child-bearing age and who does not agree to use adequate contraceptive precautions, i.e. double-barrier methods (e.g. diaphragm plus condom) or abstinence for the duration of the study and for 1 month after the last administration of the study drug,
22. Subjects who do not agree or are unable to meet the study requirements,
23. Psychological, familial, sociological or geographical conditions potentially hampering compliance with the study protocol and the follow-up schedule. Such conditions should be discussed with the patient before enrolment in the clinical trial

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
Progression-free survival at one year | 12 months after inclusion
  Percentage of subjects still alive and progression free 12 months after inclusion in the study

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 42 months
  Time (months) from inclusion in the trial until disease progression or death
Objective response rate | 42 months
  Proportion of patients with an objective response (complete or partial response) according to RECIST 1.1 criteria
Disease control rate | 42 months
  Proportion of patients with disease control (complete response, partial response or stable disease)
Duration of response | 42 months
  Time (months) from the first confirmation of objective response according to RECIST 1.1 criteria until disease progression or death
Time to response | 18 months
  Time (months) from inclusion in the trial until the date of the first confirmation of objective response according to RECIST 1.1 criteria
Overall survival (OS) | 42 months
  Time (months) from inclusion in the trial until death of the patient
Time to treatment failure | 18 months
  Time (months) from inclusion in the trial until progression, death or discontinuation due to toxicity
Proportion of patients with early tumour shrinkage (ETS) | 2 months
  Defined as tumour shrinkage ≥ 30% at the first tumour assessment based on RECIST 1.1 criteria
Depth of response (DpR) | 18 months
  Measured as the maximum reduction ratio (percentage) of the tumour compared with baseline measurement (sum of diameters of the lesions) at the different assessments based on RECIST 1.1 criteria
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 42 months
  Incidence and severity of adverse events. AEs description according to the NCI (National Cancer Institute) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03
Combined analysis of prognostic factors in metastatic disease | 42 months
  To analyse the number of lesions in liver and lung disease (1-3 vs 4-9 or ≥10), and the size of the largest lesion (<5 cm or ≥ 5 cm), in correlation with the analytical values, mainly LDH and AP values.

OTHER OUTCOMES:
RAS/BRAF conversion proportion | At treatment initiation and at the time of PD (42 months)
  Conversion rate of RAS/BRAF status at first-line treatment initiation and at the time of disease progression
RAS/BRAF mutations' detection proportion | At baseline
  Detection rate of RAS/BRAF mutations in liquid biopsies at baseline in subjects with RAS/BRAF wild-type mCRC according to the solid biopsy analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Feliu, MD, Study Director — Hospital Universitario La Paz
Locations (12):
- Spain (12):
  - ICO L´Hospitalet de Llobregat - Hospital Durán i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Sant Joan Despí-Moises Broggi, Sant Joan Despí, Barcelona
  - Hospital Universitario Puerta de Hierro-Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Rey Juan Carlos, Móstoles, Madrid
  - Hospital Clínic, Barcelona
  - Hospital General Universitario de Elda, Elda
  - Hospital Universitario Arnau de Vilanova, Lleida
  - Hospital Universitario la Paz, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario Son Espases, Palma
  - Hospital Parc Taulí, Sabadell
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: GEMCAD web page — https://www.gemcad.es/